CLINICAL TRIAL: NCT02134418
Title: Evaluation of an Intervention Program Designed to Improve Understanding of Irony on the Hemispheric Processing of Ambiguous Figurative Language in Adults With Schizophrenia
Brief Title: Evaluation of Social Skills Intervention on Cognitive Function in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0126-13-COM
Record Dates: First submitted 2014-04-30; First posted 2014-05-09 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Irony; Hemispheric processing; Theory of mind
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irony CBT training (Experimental): CBT of irony comprehension
  Interventions: Behavioral: CBT of irony comprehension
- No Intervention (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: CBT of irony comprehension — Over the course of intervention participants will analyze and discuss short film scenario's that end with an ironic statement, and will experience completing short scenario's that contain irony. Intervention will include 5 sessions, each session will take 40 minutes, 3-5 subjects will participate in each group.
  Arms: Irony CBT training

SUMMARY:
Intervention aimed at improving understanding of irony in social situations by using movies and comic strip will improve theory of mind.

DETAILED DESCRIPTION:
The overreaching goal of this study is to examine the influence of short CBT of irony comprehension on hemispheric involvement of adults with Schizophrenia. To obtain this goal a three phase study have been designed.

In the first phase all participants will be asked to fill out questionnaires screening for, cognitive abilities (TONI-3 third edition), vocabulary (Hebrew adaptation of Wechsler Adult Intelligence Scale-Third Edition, WAIS 3 HEB, Wechsler 1997), executive function capabilities and figurative language understanding (irony and metaphor) .Theory of Mind comprehension will also be assessed by using The Hinting Test (Corcoran et al.1995).

Hemispheric processing will be examined by two behavioral hemispheric experiments using split visual field paradigm. The subject sits in front of a computer screen, reads a prime sentence, and reacts to a lateralized target word.

In the first experiment- Idioms experiment, the target word in each trail would be related to the meaning of a preceding prime idiom or associated to its literal meaning .The participant is instructed to indicate as rapidly and accurately as possible whether the target word stimulus is a meaningful word or non- word. In the second experiment- irony experiment, the target word in each trail would be a literal, ironic or unrelated ending to the preceding prime sentence .Subjects would be asked to relate to the target word and to indicate as rapidly and accurately as possible whether the target word stimulus formed a meaningful expression with the preceding prime. Stimulus presentation and response would be controlled and recorded by Super-Lab 4.5 software.

The first phase will be carried out in 1-2 sessions.

In the second phase subjects will participate in a social intervention program for comprehension of verbal irony. Over the course of intervention participants will analyze and discuss short film scenario's that end with an ironic statement, and will experience completing short scenario's that contain irony. Intervention will include 5 sessions, 3-5 subjects will participate in each group.

In the third phase participants will undergo the Irony behavioral hemispheric experiment to examine changes in hemispheric processing when exposed to irony after treatment, the irony and metaphor questioners and the Hinting test. This phase will be carried out in one session.

35 subjects will participate in the study, 20 in the study group and 15 in the control group.

Subjects in the control group will watch the short film scenario's that end with an ironic statement and rank each video for its comprehensibility and their level of enjoyment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Schizophrenia
* Native Hebrew speakers
* Right handed ( subjects report)
* Without learning difficulties and who have completed 12 years of schooling (subjects report)
* Without neurological disorders ( subjects report)
* Normal or corrected to normal vision ( subjects report)

Exclusion Criteria:

* People suffering from any disabilities or handicap which limits their judgment
* With a guardian

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Irony behavioral hemispheric results | 2 months
  Changes in the response time and accuracy percentage of each hemisphere in the irony behavioral hemispheric experiment.

SECONDARY OUTCOMES:
Improved theory of mind abilities | 2 months
  The Hinting Task used to measure TOM in Schizophrenia will be used before and after the intervention (Corcoran et al.1995)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Dolfin, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Brull- Tel Aviv Community Mental Health Center, Tel Aviv, Select Your State, Israel